CLINICAL TRIAL: NCT03861312
Title: Effects of Laterality Discrimination in Patients With Non-specific Chronic Neck Pain. Randomized Blind Clinical Trial
Brief Title: Laterality Discrimination in Patients With Non-specific Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Jose Vicente Leon Hernandez, Principal Investigator, Clinical Professor, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSEULS-PI-155/2017
Record Dates: First submitted 2019-02-26; First posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Neck Pain
Keywords: Laterality task, neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck Laterality (Experimental): It was done with 20 images of necks and 4 seconds for each image in the Vanilla program of the tablet application.
  Interventions: Behavioral: Neck Laterality
- Foot Laterality (Experimental): It was done with 20 images of feet and 4 seconds for each image in the Vanilla program of the tablet application.
  Interventions: Behavioral: Foot Laterality

INTERVENTIONS:
Behavioral: Neck Laterality — Patients who belonged to the neck group performed the recognition of laterality with certain parameters. The execution of the recognition began with a test to familiarize themselves with the program at the "Basic" level and then followed the laterality test. It was done with 20 images and 4 seconds for each image in the "Vanilla" program
  Arms: Neck Laterality
Behavioral: Foot Laterality — Patients who belonged to the foot group performed the recognition of laterality with certain parameters. The execution of the recognition began with a test to familiarize themselves with the program at the "Basic" level and then followed the laterality test. It was done with 20 images and 4 seconds for each image in the "Vanilla" program
  Arms: Foot Laterality

SUMMARY:
Chronic neck pain is one of the most common causes of pain, affecting 15% of the adult population, and the fourth leading cause of disability. The recognition of laterality is the ability to recognize a part of the body that belongs to the left or right which is used as a tool to create a normal process of motor planning.

DETAILED DESCRIPTION:
The most consistent data come from the investigation of the primary motor cortex, in which the cortical representations of the altered body part are affected when there is chronic pain. Occasionally, the primary motor cortex is smaller on the affected side than on the contralateral side.

Recognition of the body schema is altered in the presence of painful disorders. The most common way of assessing the body schema is by motor imagery through the laterality discrimination of the left and right.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were as follows: a) men and women aged between 18- and 65-years b) medical diagnosis of Non-Specific Chronic Neck Pain with more than 6 months of evolution of neck pain.

Exclusion Criteria:

* Exclusion criteria included the following: a) patients with rheumatic diseases, cervical hernia, cervical whiplash syndrome, neck surgeries or history of arthrodesis, b) systemic diseases, c) vision, hearing or vestibular problems, d) Severe trauma or traffic accident which has had an impact on the cervical area.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Response time | Immediately post-intervention
  Changes in the time response. Time response is defined as the time between the image appearance and the subject response.
Accuracy | Immediately post-intervention
  Changes in the accuracy at the end of the intervention. Accuracy must be taken as the precision of the response when a subject say wether the image is right or left. It is measured by percentage of success.
Joint Position Error | Immediately post-intervention
  Changes in the joint position error at the end of the intervention. It is measured on centimeters.
Cervical Active Range of Motion | immediately post-intervention
  Changes the cervical active range of motion at the end of the intervention. It is measured on centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: David Marcos Lorenzo, Msc, Study Chair — d.marcosl20@gmail.com